CLINICAL TRIAL: NCT00944632
Title: Double-blind, Randomized, Dose Escalation Study of the Efficacy and Safety of ZK 245186 Ointment in Concentrations of 0.01%, 0.03%, and 0.1% Over 4 Weeks in Patients With Atopic Dermatitis
Brief Title: Dose Escalation of Different Concentrations of ZK 245186 in Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14501; 1402942 (Other: Company internal)
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — R-1,1,1-trifluoro-4-(5-fluoro-2,3-dihydrobenzofuran-7-yl)-4-methyl-2-(((2-methyl-5-quinolyl)amino)methyl)pentan-2-ol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Zk 245186 0.01% ointment (Active Comparator): Active treatment, lowest dose
  Interventions: Drug: ZK 245186
- ZK 245186 0.03% ointment (Active Comparator): Active comparator middle dose
  Interventions: Drug: ZK 245186
- ZK 245186 0.1% ointment (Active Comparator): Active comparator highest dose
  Interventions: Drug: ZK 245186
- Vehicle ointment (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo (vehicle ointment)

INTERVENTIONS:
Drug: ZK 245186 — Once daily topical non-occlusive application for up to 4 weeks
  Arms: ZK 245186 0.03% ointment; ZK 245186 0.1% ointment; Zk 245186 0.01% ointment
Drug: Placebo (vehicle ointment) — Once daily topical non-occlusive application for up to 4 weeks
  Arms: Vehicle ointment

SUMMARY:
The purpose of this study is to determine the safety and efficacy of three concentrations of ZK 245186 ointment and vehicle on increasing body surface areas for the treatment of atopic dermatitis and to obtain dose-response information for the three concentrations.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of atopic dermatitis (Hanifin and Rajka criteria)
* mild to moderate atopic dermatitis at beginning of study
* wash-out periods for systemic and topical treatments for atopic dermatitis
* females must use effective contraception

Exclusion Criteria:

* pregnant or lactating women
* conditions that in the opinion of the investigator may pose a risk or interfere with the evaluation of the study
* wide-spread atopic dermatitis requiring systemic treatment
* diagnosed with immunocompromised status
* skin diseases - other than atopic dermatitis - in the treatment area
* mental handicap or legally incompetent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-07-15 (Actual); Primary Completion 2010-09-15 (Actual); Study Completion 2010-09-15 (Actual)

PRIMARY OUTCOMES:
Assessment of the severity of atopic dermatitis at target lesion, based on clinical signs of inflammation | up to 4 weeks

SECONDARY OUTCOMES:
Investigator's Global Assessment of target area | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- South Africa (3):
  - PAREXEL International (Bloemfontein), Bloemfontein
  - PAREXEL International (George), George
  - PAREXEL International (Port Elizabeth), Newton Park